CLINICAL TRIAL: NCT04730791
Title: Reliability and Validity of the IASP Clinical Criteria for Identifying Patients with Nociplastic Pain
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Collaborators: KAT General Hospital (Other)
Responsible Party: Principal Investigator, Paraskevi Bilika, Study Director, University of Thessaly
Other Study IDs: 4
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Chronic Pain; Central Sensitisation; Nociplastic Pain
Keywords: Algo(s)rithm; Vignette Method; Central Sensitisation; Chronic Pain Categorization; IASP criteria; Nociplastic pain
MeSH Terms: conditions — Chronic Pain; Nociplastic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Chronic Pain Patients: Adult patients 18-65 years, with chronic pain lasting for 3 or more months, with a pain intensity of at least 3 on a 0-10 numerical pain rating scale on most days.
  Interventions: Diagnostic Test: Algo(s)rithm/ IASP clinical criteria; Diagnostic Test: Pressure Pain Threshold
- Control Group: Free pain participants
  Interventions: Diagnostic Test: Algo(s)rithm/ IASP clinical criteria; Diagnostic Test: Pressure Pain Threshold

INTERVENTIONS:
Diagnostic Test: Algo(s)rithm/ IASP clinical criteria — IASP clinical criteria for identifying nociplastic pain. The criteria is completed by the healthcare professional and includes questions about the patient's clinical picture.
Diagnostic Test: Pressure Pain Threshold — The pain pressure threshold (PPT) is used to measure pain sensitivity in body areas. The test quantifies the minimum amount of pressure in a given area, during an increasing skin pressure stimulus, which is capable of altering the feeling of pressure in pain.

SUMMARY:
This protocol will report on the validation of IASP clinical criteria for indentifying nociplastic pain. The study will include 2 phases. In the first phase, the vignette method will be used while the second phase will include the use of the algorithm in the evaluation of patients with chronic pain.

DETAILED DESCRIPTION:
For the purposes of the study, in the first phase, clinical vignettes will be created, ie short hypothetical scenarios of patients with chronic musculoskeletal pain. The vignettes will feature patients with and without nocipalstic pain. Initially, two experts will evaluate and characterize which vignettes concern patients with nociplastic pain.

Next, a team of physiotherapists with knowledge of chronic pain and CS will evaluate vignettes twice according to the IASP criteria. There will be an interval of 1 month between the two measurements. One month later, the evaluation will be repeated. The investigators will design an Android application "Algo (s) rithm" to enter the questions of the algorithm. In the second phase, Algo (s)rithm app will use to evaluate patients with chronic pain (including patients with fibromyalgia) and healthy. The investigators will compare the result with PPT measurements in the same population.In the present study the inter-rater and test-retest reliability, criterion validity, construct validity will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18-65 years
* with pain > 3months, intensity of at least 3 on a 0-10 numerical pain rating scale on most days
* or patients with fibromyalgia (according to the "criteria for classification of fibromyalgia" by the American college of rheumatology (Wolfe et al 1990)).

Exclusion Criteria:

* Patients who follow a physical therapy program
* Recent surgery or trauma
* Pregnant women,
* Patients with neurological disorders or systemic diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The measurements will be performed in the research laboratory of Clinical Exercise Physiology and Rehabilitation (CeprLab) of the University of Thessaly. The sample will consist of people who will have access to the laboratory regardless of the area of residence. The participants will be informed through the media (social networking pages, the official page of the University, the official page of the CeprLab, brochures that will be sent to physiotherapists and the Panhellenic Association of Physiotherapists).
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
IASP clinical criteria | through study completion, an average of 1 year
  IASP clinical criteria for indentifying nociplastic pain. The criteria are completed by the healthcare professional and includes questions about the patient's clinical picture.
Pressure Pain Thresholds PPT | through study completion, an average of 1 year
  The pain pressure threshold (PPT) is used to measure pain sensitivity in body areas. The test quantifies the minimum amount of pressure in a given area, during an increasing pressure of the skin, which is able to change the feeling of pressure in the pain. Measurements will be performed according to protocols used in previous studies.

CONTACTS AND LOCATIONS:
Overall Officials: Eleni V Kapreli, MSc,PhD, Study Chair — Clinical Exercise Physiology & Rehabilitation Laboratory,University of Thessaly
Locations (2):
- Greece (2):
  - Clinical Exercise Physiology and Rehabilitation Laboratory, Lamia, Central Greece
  - KAT Attica General Hospital, Athens

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smart KM, Blake C, Staines A, Doody C. The Discriminative validity of "nociceptive," "peripheral neuropathic," and "central sensitization" as mechanisms-based classifications of musculoskeletal pain. Clin J Pain. 2011 Oct;27(8):655-63. doi: 10.1097/AJP.0b013e318215f16a. PMID 21471812
- [Background] Nijs J, Apeldoorn A, Hallegraeff H, Clark J, Smeets R, Malfliet A, Girbes EL, De Kooning M, Ickmans K. Low back pain: guidelines for the clinical classification of predominant neuropathic, nociceptive, or central sensitization pain. Pain Physician. 2015 May-Jun;18(3):E333-46. PMID 26000680
- [Background] Lluch E, Nijs J, Courtney CA, Rebbeck T, Wylde V, Baert I, Wideman TH, Howells N, Skou ST. Clinical descriptors for the recognition of central sensitization pain in patients with knee osteoarthritis. Disabil Rehabil. 2018 Nov;40(23):2836-2845. doi: 10.1080/09638288.2017.1358770. Epub 2017 Aug 2. PMID 28768437
- [Background] Levesque A, Riant T, Ploteau S, Rigaud J, Labat JJ; Convergences PP Network. Clinical Criteria of Central Sensitization in Chronic Pelvic and Perineal Pain (Convergences PP Criteria): Elaboration of a Clinical Evaluation Tool Based on Formal Expert Consensus. Pain Med. 2018 Oct 1;19(10):2009-2015. doi: 10.1093/pm/pny030. PMID 29522121
- [Background] Nijs J, Leysen L, Adriaenssens N, Aguilar Ferrandiz ME, Devoogdt N, Tassenoy A, Ickmans K, Goubert D, van Wilgen CP, Wijma AJ, Kuppens K, Hoelen W, Hoelen A, Moloney N, Meeus M. Pain following cancer treatment: Guidelines for the clinical classification of predominant neuropathic, nociceptive and central sensitization pain. Acta Oncol. 2016 Jun;55(6):659-63. doi: 10.3109/0284186X.2016.1167958. Epub 2016 May 4. PMID 27142228
- [Background] Nijs J, Polli A, Willaert W, Malfliet A, Huysmans E, Coppieters I. Central sensitisation: another label or useful diagnosis? Drug Ther Bull. 2019 Apr;57(4):60-63. doi: 10.1136/dtb.2018.000035. Epub 2019 Mar 11. No abstract available. PMID 30858291
- [Background] Smart KM, Blake C, Staines A, Thacker M, Doody C. Mechanisms-based classifications of musculoskeletal pain: part 1 of 3: symptoms and signs of central sensitisation in patients with low back (+/- leg) pain. Man Ther. 2012 Aug;17(4):336-44. doi: 10.1016/j.math.2012.03.013. Epub 2012 Apr 23. PMID 22534654
- [Background] Stacey D, Briere N, Robitaille H, Fraser K, Desroches S, Legare F. A systematic process for creating and appraising clinical vignettes to illustrate interprofessional shared decision making. J Interprof Care. 2014 Sep;28(5):453-9. doi: 10.3109/13561820.2014.911157. Epub 2014 Apr 28. PMID 24766619
- [Background] Nijs J, Lahousse A, Kapreli E, Bilika P, Saracoglu I, Malfliet A, Coppieters I, De Baets L, Leysen L, Roose E, Clark J, Voogt L, Huysmans E. Nociplastic Pain Criteria or Recognition of Central Sensitization? Pain Phenotyping in the Past, Present and Future. J Clin Med. 2021 Jul 21;10(15):3203. doi: 10.3390/jcm10153203. PMID 34361986
- [Background] Kosek E, Clauw D, Nijs J, Baron R, Gilron I, Harris RE, Mico JA, Rice ASC, Sterling M. Chronic nociplastic pain affecting the musculoskeletal system: clinical criteria and grading system. Pain. 2021 Nov 1;162(11):2629-2634. doi: 10.1097/j.pain.0000000000002324. No abstract available. PMID 33974577